CLINICAL TRIAL: NCT04457726
Title: Part Two of Novel Adoptive Cellular Therapy With SARS-CoV-2 Specific T Cells in Patients With Severe COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Duke-NUS Graduate Medical School (Other); National University Hospital, Singapore (Other); Singapore General Hospital (Other); Sengkang General Hospital (Other); Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-T 2.0
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recipients with severe COVID-19 (Experimental): Recipients who are confirmed positive by SARS-CoV-2 testing and have severe COVID-19.
  Interventions: Biological: SARS-CoV-2 Specific T Cells
- Recipients with mild to moderate COVID-19 (Experimental): Recipients who are confirmed positive by SARS-CoV-2 testing and have mild to moderate COVID-19.
  Interventions: Biological: SARS-CoV-2 Specific T Cells

INTERVENTIONS:
Biological: SARS-CoV-2 Specific T Cells — Eligible patients will receive a single infusion of SARS-CoV-2 specific T cells intravenously.

SUMMARY:
The overall objective of this project is to develop an emergent treatment protocol using adoptive T-cell therapy for the treatment of severe COVID-19. The central hypothesis is that SARS-CoV-2 specific T cells from convalescent donors who have recovered from COVID-19 can be manufactured expeditiously and these cells are safe and effective for the treatment of severe SARS-CoV-2 infections.

DETAILED DESCRIPTION:
A novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the cause of Coronavirus Disease 2019 (COVID-19). Currently, no vaccine has been proven to be effective. While waiting for vaccine to be developed, passive immunity can be acquired immediately by adoptive transfer of SARS-CoV-2 specific T cells from convalescent donors into newly infected patients.

The overall objective of this project is to develop an emergent treatment protocol using adoptive T-cell therapy for the treatment of severe COVID-19. The central hypothesis is that SARS-CoV-2 specific T cells from convalescent donors who have recovered from COVID-19 can be manufactured expeditiously and these cells are safe and effective for the treatment of severe SARS-CoV-2 infections. Part Two of this project is to assess the safety and efficacy of these T cells in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to 90 years
* Tested positive for SARS-CoV-2 <72 hours prior to enrolment
* Predicted to have high chance of mortality:

Group 1: Severe disease, defined by one or more of the following:

* Dyspnea
* Respiratory frequency ≥ 30/min
* Blood oxygen saturation ≤ 93%
* Partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300
* Lung infiltrates > 50% within 24 to 48 hours
* Respiratory failure
* Septic shock
* Multiple organ dysfunction or failure

Group 2: Mild to moderate disease, at high risk of progression to severe disease. For example,

* Age > 65 years
* Chronic health conditions such as chronic lung disease, cardiovascular disease, diabetes mellitus, obesity, end-stage renal disease or liver disease

Exclusion Criteria:

* Rapidly progressive disease with anticipated life-expectancy <72 hours
* Receiving steroid (>0.5mg/kg methylprednisolone equivalent)
* Pregnancy
* Breastfeeding

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities | till Day 28 after infusion of SARS-CoV-2 specific T cells
  Dose-limiting toxicities are defined as >Grade 3 Common Toxicity Criteria associated with the therapeutic cells. Toxicity rate will be summarized descriptively.

SECONDARY OUTCOMES:
National Early Warning Score (NEWS) | one month
  Measured by change in daily NEWS score after infusion of SARS-CoV-2 specific T cells
Time to improvement by one category on a WHO ordinal scale | one month
  Measured by time-to-improvement by one category on a WHO ordinal scale after infusion of SARS-CoV-2 specific T cells
Time-to-SARS-CoV-2 negativity after infusion of SARS-CoV-2 specific T cells | two months
  Measured by time-to-SARS-CoV-2 negativity after infusion of SARS-CoV-2 specific T cells
Duration of persistence of SARS-CoV-2 specific T cells in the recipient's blood circulation | two months
  Measured by the duration of persistence of SARS-CoV-2 specific T cells in the recipient's blood
Time-to-normalization of cytokine level, lymphocyte subsets, and gene transcriptome after T cell infusion | two months
  Measured by the time-to-normalization of cytokine level, lymphocyte subsets, and gene transcriptome after T cell infusion
Overall survival (OS) at 3 months after infusion of SARS-CoV-2 specific T cells | three months
  Measured by the proportion of recipients surviving at 3 months after infusion of SARS-CoV-2 specific T cells

CONTACTS AND LOCATIONS:
Overall Officials: Wing Hang Leung, Principal Investigator — KK Hospital, SingHealth Duke NUS
Locations (5):
- Singapore (5):
  - Changi General Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
  - National University Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - Singapore General Hospital, Singapore